CLINICAL TRIAL: NCT07096895
Title: EUS-directed Transenteric ERCP (EDEE) in Patients With Benign and Malignant Underlying Conditions and Inaccessible Papilla/Biliodigestive Anastomosis (BDA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelisches Krankenhaus Düsseldorf (Other)
Responsible Party: Principal Investigator, Torsten Beyna, PD Dr. med, Evangelisches Krankenhaus Düsseldorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDEE EVK Duesseldorf
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Biliary Intervention; Altered Anatomy; Malignant Gastric Outlet Obstruction; EUS Guided Enteroenteric Anastomosis; EDEE
Keywords: ERCP; altered anatomy; EUS; anastomosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EDEE (Experimental)
  Interventions: Procedure: EDEE (EUS-directed transenteric ERCP)

INTERVENTIONS:
Procedure: EDEE (EUS-directed transenteric ERCP) — Technical aspects of EUS-guided anastomosis and ERCP via LAMS (Lumen apposing metal stent)

SUMMARY:
Safety and efficacy of EDEE (EUS-directed transenteric ERCP)

DETAILED DESCRIPTION:
Background and Study Objective Endoscopic retrograde cholangiopancreatography (ERCP) is considered the gold standard when biliary intervention is indicated. However, there are situations where conventional ERCP is no longer feasible - for example, in the presence of malignant gastric outlet obstruction.

Additionally, the number of patients with surgically altered anatomy due to benign or malignant underlying diseases is increasing. For this group of patients, enteroscopy-assisted ERCP can generally be considered. However, the success rate of this procedure varies depending on the anatomical situation and is only around 61.7%. Therefore, patients in whom the papilla or the biliodigestive anastomosis (BDA) cannot be reached either via conventional endoscopy or enteroscopy-assisted ERCP - yet require biliary intervention - present a particular clinical challenge.

Traditionally, the only option in such cases has often been percutaneous transhepatic drainage (PTBD). This approach frequently requires repeated procedures over several months and, in some cases, results in a permanent external drainage. In recent years, endoscopic ultrasound (EUS)-guided techniques have emerged as a promising treatment option for this patient population. These methods show a high technical success rate of approximately 90%, but are not suitable in cases requiring complex interventions (e.g., multiple strictures of the BDA) or when targeting the right biliary system.

An alternative approach involves a two-step procedure: first, an EUS-guided entero-enteric anastomosis is created using a lumen-apposing metal stent (LAMS); in a second step, ERCP is performed via the LAMS. This procedure is referred to in the literature as Endoscopic Ultrasound-Directed Transenteric ERCP (EDEE).

Since only a few systematic studies on this alternative procedure have been published so far, the objective of this retrospective study is to assess the technical and clinical success rates and evaluate the safety of EDEE.

ELIGIBILITY:
Inclusion Criteria:

* signed consent form
* Indication for an EDEE
* Age >18 years

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | during the procedure
  number an rate of patients with successful creation of gastro-enterostomy followed by successfull ERCP via LAMS (lumen apposing metal stent) including all planned interventions
Safety of EDEE | during the procedure
  number and rate of patients, in whom a procedure related complication occured

SECONDARY OUTCOMES:
Clinical success rate | at the day of last procedure
  absence of need for alternative drainage
Technical aspects of gastro-enterostomy | during the procedure
  Evaluation of devices and potential pitfalls creating a gastroenterostomy
Techinical aspect of ERCP via LAMS | during procedure
  Evaluation of devices and potential pitfalls performing ERCP via LAMS
Requirement for reinterventions | during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Torsten PD Dr. med Beyna, Principal Investigator — Evangelisches Krankenhaus Düsseldorf
Locations (1):
- Evangelisches Krankenhaus Düsseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No